CLINICAL TRIAL: NCT04573452
Title: The Role of Galectin-3 in the Pathogenesis and Prediction of Placenta Accreta
Brief Title: Galectin-3 and Placenta Accreta
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Other Study IDs: G-PA
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal pregnancy group
  Interventions: Diagnostic Test: Galectin-3; Diagnostic Test: Placental Galactin-3
- Placenta accreta at 24-32 weeks group
  Interventions: Diagnostic Test: Galectin-3; Diagnostic Test: Placental Galactin-3

INTERVENTIONS:
Diagnostic Test: Galectin-3 — Measurement of Gal-3 in Serum which will be isolated from the blood samples by ELISA (Enzyme-Linked immunosorbent Assay) (R&D Systems, Minneapolis, MN, USA).
Diagnostic Test: Placental Galactin-3 — Measurement of Gal-3 in Villous and decidual tissues homogenate by ELISA

SUMMARY:
Galectins are a family of carbohydrate-binding proteins that have a high affinity to galactosides, its protein portion is located in the nucleus and the cytoplasm with its carbohydrate recognition domain which has high ability to be glycosylated inside or outside the cell.

They are expressed by vascular endothelium, immune cells (macrophages, neutrophils, and mast cells), uterus, placenta, cardiac muscle, liver, epithelium of the gastrointestinal tract, and many other tissues.

Although some galectins have intracellular functions, the majority of them have extracellular activities, which facilitate their contribution to cell adhesion, cell activation, and inflammation. Galectin-3 (Gal-3) is a unique pentamer of the galectins family and it is involved in both physiological functions; cell growth and differentiation, and pathological conditions; inflammation, fibrosis, and metastasis.

Regarding pregnancy, Gal-3 is proved to participate in angiogenesis, embryo developmental processes, and modulation of maternal immunity.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 28-32 weeks.
2. Age between 20-40 years.
3. Singleton pregnancy.
4. Women with suspicion of placenta accreta
5. Cases with mild vaginal bleeding or not having any vaginal bleeding.

Exclusion Criteria:

1. Women are known to have any medical disorders.
2. Patients with known bleeding disorders or on anticoagulant therapy.
3. Patients refuse to participate.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Galactin 3 level in the blood | 6 weeks
  measured by ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt